CLINICAL TRIAL: NCT01382680
Title: Comparison of the Use of the Guide-wire G-240 to a Combination of a Flexible/Hydrophil Guide Wire With a Nitinol Wire in Patients With Stenosis of the Bile Ducts in ERCP
Brief Title: Comparison of the Guide-wire G-240 to a Combination of a Flexible/Hydrophil and a Nitinol Guide Wire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Jorg Albert, Johann Wolfgang Goethe-University Hospitals, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 136/10
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Other Specified Diseases of Biliary Tract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Classic guidewires (Active Comparator): Conventional guidewires used in combination as preferred by the investigating ERCP specialist
  Interventions: Device: Guidewire
- New guidewire (G240) (Active Comparator): Primary use of the new guidewire (G240)
  Interventions: Device: Guidewire

INTERVENTIONS:
Device: Guidewire — Use of a guidewire at ERCP for cannulating a stenosis of the biliary tract and for applying a therapeutic device (stent, dilation catheter, others)
  Other Names: Terumo; RF-GA25263M, RF-GS25263M, RF-GS32403M, RF-PS25453M; G-240 2527S/A, G-240 2545S/A, G-240 3527S/A, G-240 545S/A

SUMMARY:
In ERCP practice, most often a combined use of guidewires is necessary to attain a therapeutic aim. E.g. a hyperflexible hydrophilic guidewire is changed after cannulating a stricture to a nitinol wire for improved stability with the use of therapeutic devices. A new guide-wire (G240) combines these characteristics with a stable shaft and a hydrophilic tip. The investigators test the hypothesis that the use of this new guidewire would decrease number of guidewires used within one ERCP session.

DETAILED DESCRIPTION:
This is a randomized, monocentric study.

ELIGIBILITY:
Inclusion Criteria:

* Obstruction of the biliary tract (cross sectional imaging or ultrasonography/lab data)

Exclusion Criteria:

* Operatively alternated anatomy of the patient.
* Intervention of the pancreatic duct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of guidewires per ERCP session | Within the same ERCP session (day 1)

SECONDARY OUTCOMES:
Treatment aim | day 1
  Comparison of number of patients in whom the treatment aim could be achieved in both study groups
Time of ERCP session | day 1
  Comparison of time needed for the ERCP session in both study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg G Albert, MD, Principal Investigator — Johann Wolfgang Goethe University Hospital and Clinics Department of Internal Medicine I
Locations (1):
- Department of Internal Medicine I, Frankfurt, Germany

REFERENCES:
- [Derived] Albert JG, Lucas K, Filmann N, Herrmann E, Schroder O, Sarrazin C, Trojan J, Kronenberger B, Bojunga J, Zeuzem S, Friedrich-Rust M. A novel, stiff-shaft, flexible-tip guidewire for cannulation of biliary stricture during endoscopic retrograde cholangiopancreatography: a randomized trial. Endoscopy. 2014 Oct;46(10):857-61. doi: 10.1055/s-0034-1377628. Epub 2014 Sep 10. PMID 25208030